CLINICAL TRIAL: NCT05310136
Title: Effects of Nurse-led Brief Behavioral Treatment for Insomnia: A Feasibility Randomized Controlled Trial
Brief Title: Nurse-led BBTI for Improving Insomnia Severity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202111028
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
Keywords: BBTI; adult
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nurse-guided BBTi intervention group (Experimental): Participants will experience 4-week treatment period (2 in person and 2 via telephone).
  Interventions: Behavioral: BBTi
- Control group (No Intervention): Participants will received sleep hygiene at the enrollment of the study and be required to maintain their usual lifestyle and medical treatment for 4 weeks.

INTERVENTIONS:
Behavioral: BBTi — On the arrival for the baseline appointment, participants will receive workbooks which include an outline and content of BBTi, sleep diaries, and adherence record. In the end of weeks 1 and 3, nurse interventionist will meet participants to review their sleep diary data and negotiate their bedtime and wake-time schedule. During the weeks 2 and 4, participants will receive planned follow-up phone calls to assess their adherence and review progress and challenges.
  Arms: Nurse-guided BBTi intervention group

SUMMARY:
Brief behavioral treatment for insomnia (BBTI) is a new treatment direction for primary and comorbid insomnia; however, its treatment model has not been established in Taiwan. This study aims to establish the BBTI treatment model among insomniacs in Taiwan and to examine the immediate effects of nurse-led BBTI in adults with insomnia complaints. In this assessor-blinded randomized controlled trial, participants will be randomly allocated to the nurse-led BBTI experimental group, or sleep hygiene control group. Measurement outcomes are sleep parameters measured by the Chinese version of Insomnia Severity Index, Chinese version of Pittsburgh sleep quality index, and sleep diary. Questionnaires will be assessed in pretreatment, posttreatment, and one-month follow-up. We hypothesize that adults with insomnia complaints undergoing nurse-led BBTI will experience greater alleviations in sleep in comparison with participants in the sleep hygiene control group.

DETAILED DESCRIPTION:
Background: Insomnia, defined as difficulty initiating and maintaining sleep such that it interferes with daytime function, is a common complaint among the general population, which in turn undermine their mood, cognitive functions, and quality of life. Brief behavioral treatment for insomnia (BBTI) is a new treatment direction for primary and comorbid insomnia; however, its treatment model has not been established in Taiwan.

Purposes: To establish the BBTi treatment model among insomniacs in Taiwan and to examine the immediate effects of nurse-led BBTI in adults with insomnia complaints. We hypothesize that adults with insomnia complaints undergoing nurse-led BBTI will experience greater alleviations in sleep in comparison with participants in the sleep hygiene control group.

Methods: This assessor-blinded randomized controlled trial will employ a two-arm parallel-group design. A total of 42 adults with insomnia complaints will be randomly allocated to the nurse-led BBTI, or sleep hygiene control group in a 1:1 ratio. For the nurse-led BBTI group, all participants will experience 4-week nurse-led BBTi via 2 in person and 2 telephone sessions. The contents include sleep hygiene, stimulus control, sleep restriction, and relaxation. For the sleep hygiene control group, they will receive usual care, sleep hygiene education, and weekly LINE contacts. Measurement outcomes are sleep parameters measured by the Chinese version of Insomnia Severity Index, Chinese version of Pittsburgh sleep quality index, and sleep diary. Questionnaires will be assessed in pretreatment, posttreatment, and one-month follow-up. A generalized estimating equation will be used to test research hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. Report lying awake for ≥30 min a night for ≥3 nights per week for ≥3 months
2. Have insomnia with a total score ≥ 8 on the Chinese version of the insomnia severity index (CISI) at screening
3. Be able to communicate in Mandarin Chinese

Exclusion Criteria:

1. Premorbid diagnoses of seizure, other sleep disorders (e.g., sleep apnea, screened by using the STOP-Bang questionnaire with a score > 3), psychiatric diseases, substance abuse, and alcoholism
2. Shift workers
3. Women who are pregnant, breastfeeding, or in the menopausal transition

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in Sleep parameters from sleep logs: sleep onset latency(SOL) | At baseline, week 1 to 3 (during the intervention), and one month (follow-up)
  Sleep onset latency(SOL) is the time of duration from lying on bed to fall asleep. SOL shorter than 30 minutes is one of criteria of good sleep condition.
Changes in Sleep parameters from sleep logs: after sleep onset(WASO) | At baseline, week 1 to 3 (during the intervention), and one month (follow-up)
  Wake after sleep onset(WASO) is the total time of wakefulness after sleep onset. WASO less than 30 minutes is one of criteria of good sleep condition.
Changes in Sleep parameters from sleep logs: total sleep time(TST) | At baseline, week 1 to 3 (during the intervention), and one month (follow-up)
  Total sleep time(TST) is the total time of falling asleep. TST will be used to calculate sleep efficiency(SE).
Changes in Sleep parameters from sleep logs: sleep efficiency(SE) | At baseline, week 1 to 3 (during the intervention), and one month (follow-up)
  Sleep efficiency(SE) is the percentage of total sleep time to time in bed. A good sleep condition should meet the criteria of SE greater than 85%.
Changes in Insomnia Severity | At baseline, week 5 (after the intervention), and one month (follow-up)
  Insomnia Severity will be measured by Chinese version Insomnia Severity Index (ISI). ISI has 7 questions to evaluate sleep difficulty. The total score range from 0-28, if score>7 is associated with insomnia. The higher score means more severe insomnia.
Changes in Sleep quality | At baseline, week 5 (after the intervention), and one month (follow-up)
  Sleep quality will be measured by Pittsburgh Sleep Quality Index (PSQI). PSQI has 18 questions to evaluate sleep condition. The total score range from 0-21, if score>5 is associated with poor sleep. The higher score means poorer sleep quality.

SECONDARY OUTCOMES:
Changes in Quality of life | At baseline, week 5 (after the intervention), and one month (follow-up)
  Quality of life will be measured by RAND-36 Health Status Inventory. It has 36 questions to assess eight health concepts including physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions.
Changes in Daytime Sleepiness | At baseline, week 5 (after the intervention), and one month (follow-up)
  Daytime Sleepiness will be measured by Epworth Sleepiness Scale (ESS). ESS has 8 questions to evaluate the condition of dozing off or falling asleep. The total score range from 0-24, if score>10 is associated with daytime sleepiness.
Changes in Depression | At baseline, week 5 (after the intervention), and one month (follow-up)
  Depression will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of depression. The total score should be multiplied by 2 range from 0-42, if score>9 is associated with depression. The higher score means more severe depression.
Changes in Anxiety | At baseline, week 5 (after the intervention), and one month (follow-up)
  Anxiety will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of anxiety. The total score should be multiplied by 2 range from 0-42, if score>7 is associated with anxiety. The higher score means more severe anxiety.
Changes in Stress | At baseline, week 5 (after the intervention), and one month (follow-up)
  Stress will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of stress. The total score should be multiplied by 2 range from 0-42, if score>14 is associated with anxiety. The higher score means more severe stress.
Changes in Fatigue | At baseline, week 5 (after the intervention), and one month (follow-up)
  Stress will be measured by Brief Fatigue Inventory- Taiwan Form (BFI- Taiwan Form). BFI- Taiwan Form has 9 questions to evaluate the state of fatigue. The score of each item range from 0-10, if score>4 is associated with fatigue. The higher score means more severe fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasan F, Prasetya EC, Gordon CJ, Romadlon DS, Chang KM, Bartlett DJ, Lin CJ, Gautama MSN, Izzati N, Chiu HY. Effects of nurse-led, web-based brief behavioral therapy on insomnia severity in patients in the chronic stage of stroke recovery: a preliminary randomized controlled trial. J Clin Sleep Med. 2025 Dec 1;21(12):2031-2040. doi: 10.5664/jcsm.11856. PMID 40904277
- [Derived] Chang KM, Lin CJ, Jan YW, Gordon CJ, Lee HC, Shih CY, Bartlett DJ, Fan YC, Chiu HY. Effects of nurse-led brief behavioral treatment for insomnia in adults: a randomized controlled trial. J Clin Sleep Med. 2024 Nov 1;20(11):1763-1772. doi: 10.5664/jcsm.11256. PMID 38935053